CLINICAL TRIAL: NCT03048890
Title: VascTrac PAD ResearchKit Study
Brief Title: VascTrac Peripheral Arterial Disease (PAD) Study
Acronym: VascTrac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: W.L.Gore & Associates (Industry); Abbott (Industry); Cook Group Incorporated (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Oliver Aalami, Principal Investigator, Palo Alto Veterans Institute for Research
Other Study IDs: AAL0001ARG
Record Dates: First submitted 2016-09-06; First posted 2017-02-09 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Artery Disease; Intermittent Claudication
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with PAD: Patients with PAD will be in 1 cohort and will have their physical activity levels closely monitored by researchers and physicians.
  Interventions: Behavioral: Physical activity levels
- Patients without PAD: Patients without PAD will be allowed to contribute their data to the application, but they will not be as closely monitored.
  Interventions: Behavioral: Physical activity levels

INTERVENTIONS:
Behavioral: Physical activity levels — Patients with severely low physical activity levels will be notified to consult their physician.

SUMMARY:
VascTrac is a mobile medical application that tracks users' physical activity levels in order to predict endovascular failure of patients with Peripheral Artery Disease.

DETAILED DESCRIPTION:
VascTrac uses open-source software from Apple's ResearchKit to passively track physical activity levels of users who sign up. The goal is to predict post-intervention endovascular failure before it occurs. Currently, physicians have no way of knowing when procedures such as angioplasties fail; with VascTrac, researchers hope to find downward trends in physical activity that will predict and indicate endovascular failure. All users are assigned numbers and their medical data is securely coded, decreasing the risk of promulgation of personal information.

ELIGIBILITY:
Inclusion Criteria:

* adult, has iPhone 5s, can read English

Exclusion Criteria:

* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults with an iPhone 5s or higher who can read English
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Two Years
  Participants will have their physical activity measured and recorded by the devices in Apple's Health application.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver O Aalami, MD, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
If users consent, their data may or may not be shared with their personal physicians for direct patient care.

REFERENCES:
- [Background] Cunningham MA, Swanson V, Pappas E, O'Carroll RE, Holdsworth RJ. Illness beliefs and walking behavior after revascularization for intermittent claudication: a qualitative study. J Cardiopulm Rehabil Prev. 2014 May-Jun;34(3):195-201. doi: 10.1097/HCR.0000000000000046. PMID 24603143
- [Background] Carter T, O'Neill S, Johns N, Brady RR. Contemporary vascular smartphone medical applications. Ann Vasc Surg. 2013 Aug;27(6):804-9. doi: 10.1016/j.avsg.2012.10.013. Epub 2013 Mar 25. PMID 23535521
- [Background] Coughlin PA, Kent PJ, Turton EP, Byrne P, Berridge DC, Scott DJ, Kester RC. A new device for the measurement of disease severity in patients with intermittent claudication. Eur J Vasc Endovasc Surg. 2001 Dec;22(6):516-22. doi: 10.1053/ejvs.2001.1528. PMID 11735200
- [Background] Gernigon M, Le Faucheur A, Fradin D, Noury-Desvaux B, Landron C, Mahe G, Abraham P. Global positioning system use in the community to evaluate improvements in walking after revascularization: a prospective multicenter study with 6-month follow-up in patients with peripheral arterial disease. Medicine (Baltimore). 2015 May;94(18):e838. doi: 10.1097/MD.0000000000000838. PMID 25950694
- [Background] Afaq A, Patel JH, Gardner AW, Hennebry TA. Predictors of change in walking distance in patients with peripheral arterial disease undergoing endovascular intervention. Clin Cardiol. 2009 Sep;32(9):E7-11. doi: 10.1002/clc.20553. PMID 19645033
- [Background] Malgor RD, Alahdab F, Elraiyah TA, Rizvi AZ, Lane MA, Prokop LJ, Phung OJ, Farah W, Montori VM, Conte MS, Murad MH. A systematic review of treatment of intermittent claudication in the lower extremities. J Vasc Surg. 2015 Mar;61(3 Suppl):54S-73S. doi: 10.1016/j.jvs.2014.12.007. Epub 2015 Feb 23. PMID 25721067
- [Background] Murphy TP, Hirsch AT, Ricotta JJ, Cutlip DE, Mohler E, Regensteiner JG, Comerota AJ, Cohen DJ; CLEVER Steering Committee. The Claudication: Exercise Vs. Endoluminal Revascularization (CLEVER) study: rationale and methods. J Vasc Surg. 2008 Jun;47(6):1356-63. doi: 10.1016/j.jvs.2007.12.048. Epub 2008 Apr 25. PMID 18440181
- [Background] Murphy TP, Cutlip DE, Regensteiner JG, Mohler ER, Cohen DJ, Reynolds MR, Massaro JM, Lewis BA, Cerezo J, Oldenburg NC, Thum CC, Goldberg S, Jaff MR, Steffes MW, Comerota AJ, Ehrman J, Treat-Jacobson D, Walsh ME, Collins T, Badenhop DT, Bronas U, Hirsch AT; CLEVER Study Investigators. Supervised exercise versus primary stenting for claudication resulting from aortoiliac peripheral artery disease: six-month outcomes from the claudication: exercise versus endoluminal revascularization (CLEVER) study. Circulation. 2012 Jan 3;125(1):130-9. doi: 10.1161/CIRCULATIONAHA.111.075770. Epub 2011 Nov 16. PMID 22090168
- [Background] Murphy TP, Hirsch AT, Cutlip DE, Regensteiner JG, Comerota AJ, Mohler E, Cohen DJ, Massaro J; CLEVER Investigators. Claudication: exercise vs endoluminal revascularization (CLEVER) study update. J Vasc Surg. 2009 Oct;50(4):942-945.e2. doi: 10.1016/j.jvs.2009.04.076. Epub 2009 Aug 5. PMID 19660897